CLINICAL TRIAL: NCT02993705
Title: Phase II Trial On Trabectedin In The Treatment Of Advanced Uterine And Ovarian Carcinosarcoma (CS)
Brief Title: Trial On Trabectedin In The Treatment Of Advanced Uterine And Ovarian Carcinosarcoma (CS)
Acronym: MITO 26
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1561
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Carcinosarcoma, Ovarian; Carcinosarcomas Uterine
MeSH Terms: conditions — Carcinosarcoma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trabectedin (Experimental): Trabectedin will be infused at the dose of 1.3 mg/m2 as a 3- hour iv infusion every 3 weeks via a central venous catheter.
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Chemotherapy drug
  Other Names: Yondelis

SUMMARY:
Multicenter phase II study on trabectedin in patients advanced uterine and ovarian carcinosarcoma. Patients will receive trabectedin until disease progression or unacceptable toxicity. Disease response evaluation will be assessed every 9 weeks.

DETAILED DESCRIPTION:
This is a Phase II, multi-centre, single arm study aiming at evaluating efficacy and toxicity of Trabectedin in a population of advanced or recurrent ovarian and uterine carcinosarcoma.

Trabectedin will be infused at the dose of 1.3 mg/m2 as a 3- hour iv infusion every 3 weeks via a central venous catheter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented Stage I-IV or recurrent uterine or ovarian carcinosarcoma not amenable to surgery or radiotherapy
* No more than 2 previous chemotherapy lines
* PS 0-2 (ECOG)
* Age> 18
* Measurable disease
* Life expectancy of at least 3 months
* Adequate organ functions:

  * Hematopoietic; Absolute neutrophil count ≥ 1,500/mm^3; Platelet count ≥ 100,000/mm^3; Hemoglobin ≥ 9 g/dL Hepatic; AST and ALT ≤ 1.5 times upper limit of normal (ULN)*; Protocol Version 1.0_05.09.2016 6 Alkaline phosphatase ≤ 2.5 times ULN*; Bilirubin ≤ 1.5 times ULN NOTE: * ≤ 3 times ULN if liver metastases are present Renal; Creatinine Clearance ≥ 45 mL/min or Serum Creatinine ≤1.5 x ULN Serum Albumin >3.0 g/dL
* Previous Brachytherapy treatment for uterine carcinosarcoma is allowed
* No other invasive malignancy within the past 3 years except non-melanoma skin cancer
* Written Informed Consent

Exclusion Criteria:

* More than 2 previous chemotherapy lines
* Single tumor lesion inside a previous irradiated filed
* Pregnant (potentially fertile patients must be not in pregnancy during and for at least 3 months after study participation and must have a negative serum pregnancy test)
* Active infection requiring antibiotics
* Symptomatic peripheral neuropathy > grade 2 according to the NCI Common Toxicity Criteria.
* Congestive heart failure or angina pectoris even if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled high risk hypertension or arrhythmia.
* Unstable or severe intercurrent medical condition that, in the opinion of the investigator, might interfere with achievement of study objectives
* Psychological or sociological conditions, addictive disorders, or family problems, which would preclude compliance with the protocol

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | three years
  The primary endpoint of this study is to evaluate the activity of trabectedin in terms of the objective response rate (ORR) in patients with advanced uterine and ovarian carcinosarcoma.

SECONDARY OUTCOMES:
Duration of response | three years
Progression Free Survival (PFS) | three years
  the diagnosis of progression will be assessed by radiological criteria; CA 125 increases alone (GCIG criteria of progression) will not be considered as progression of disease without a radiological confirmation of progression
Overall Survival (OS) | three years
Adverse events | three years
  Incidence of adverse events, according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) v 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Lorusso, Prof., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoffski P, Casali PP, Taron M, et al. Impact of the DNA repair functionality on the outcome of sarcoma patients treated with trabectedin (ET-743). J Clin Oncol, 2006; 24 (18 Suppl):525s (Abstract#9522)
- [Result] Berton-Rigaud D, Devouassoux-Shisheboran M, Ledermann JA, Leitao MM, Powell MA, Poveda A, Beale P, Glasspool RM, Creutzberg CL, Harter P, Kim JW, Reed NS, Ray-Coquard I. Gynecologic Cancer InterGroup (GCIG) consensus review for uterine and ovarian carcinosarcoma. Int J Gynecol Cancer. 2014 Nov;24(9 Suppl 3):S55-60. doi: 10.1097/IGC.0000000000000228. PMID 25341582
- [Result] Makker V, Abu-Rustum NR, Alektiar KM, Aghajanian CA, Zhou Q, Iasonos A, Hensley ML. A retrospective assessment of outcomes of chemotherapy-based versus radiation-only adjuvant treatment for completely resected stage I-IV uterine carcinosarcoma. Gynecol Oncol. 2008 Nov;111(2):249-54. doi: 10.1016/j.ygyno.2008.06.035. Epub 2008 Aug 27. PMID 18755503
- [Result] Cicin I, Saip P, Eralp Y, Selam M, Topuz S, Ozluk Y, Aydin Y, Topuz E. Ovarian carcinosarcomas: clinicopathological prognostic factors and evaluation of chemotherapy regimens containing platinum. Gynecol Oncol. 2008 Jan;108(1):136-40. doi: 10.1016/j.ygyno.2007.09.003. Epub 2007 Oct 23. PMID 17936342
- [Result] Jonson AL, Bliss RL, Truskinovsky A, Judson P, Argenta P, Carson L, Dusenbery K, Downs LS Jr. Clinical features and outcomes of uterine and ovarian carcinosarcoma. Gynecol Oncol. 2006 Mar;100(3):561-4. doi: 10.1016/j.ygyno.2005.09.017. Epub 2005 Nov 4. PMID 16271748
- [Result] Reed NS, Mangioni C, Malmstrom H, Scarfone G, Poveda A, Pecorelli S, Tateo S, Franchi M, Jobsen JJ, Coens C, Teodorovic I, Vergote I, Vermorken JB; European Organisation for Research and Treatment of Cancer Gynaecological Cancer Group. Phase III randomised study to evaluate the role of adjuvant pelvic radiotherapy in the treatment of uterine sarcomas stages I and II: an European Organisation for Research and Treatment of Cancer Gynaecological Cancer Group Study (protocol 55874). Eur J Cancer. 2008 Apr;44(6):808-18. doi: 10.1016/j.ejca.2008.01.019. Epub 2008 Apr 2. PMID 18378136
- [Result] Wolfson AH, Brady MF, Rocereto T, Mannel RS, Lee YC, Futoran RJ, Cohn DE, Ioffe OB. A gynecologic oncology group randomized phase III trial of whole abdominal irradiation (WAI) vs. cisplatin-ifosfamide and mesna (CIM) as post-surgical therapy in stage I-IV carcinosarcoma (CS) of the uterus. Gynecol Oncol. 2007 Nov;107(2):177-85. doi: 10.1016/j.ygyno.2007.07.070. Epub 2007 Sep 5. PMID 17822748
- [Result] Sutton G, Brunetto VL, Kilgore L, Soper JT, McGehee R, Olt G, Lentz SS, Sorosky J, Hsiu JG. A phase III trial of ifosfamide with or without cisplatin in carcinosarcoma of the uterus: A Gynecologic Oncology Group Study. Gynecol Oncol. 2000 Nov;79(2):147-53. doi: 10.1006/gyno.2000.6001. PMID 11063636
- [Result] Sutton G, Kauderer J, Carson LF, Lentz SS, Whitney CW, Gallion H; Gynecologic Oncology Group. Adjuvant ifosfamide and cisplatin in patients with completely resected stage I or II carcinosarcomas (mixed mesodermal tumors) of the uterus: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Mar;96(3):630-4. doi: 10.1016/j.ygyno.2004.11.022. PMID 15721404
- [Result] Toyoshima M, Akahira J, Matsunaga G, Niikura H, Ito K, Yaegashi N, Tase T. Clinical experience with combination paclitaxel and carboplatin therapy for advanced or recurrent carcinosarcoma of the uterus. Gynecol Oncol. 2004 Sep;94(3):774-8. doi: 10.1016/j.ygyno.2004.05.048. PMID 15350372
- [Result] Leiser AL, Chi DS, Ishill NM, Tew WP. Carcinosarcoma of the ovary treated with platinum and taxane: the memorial Sloan-Kettering Cancer Center experience. Gynecol Oncol. 2007 Jun;105(3):657-61. doi: 10.1016/j.ygyno.2007.01.037. Epub 2007 Mar 28. PMID 17395252
- [Result] Homesley HD, Filiaci V, Markman M, Bitterman P, Eaton L, Kilgore LC, Monk BJ, Ueland FR; Gynecologic Oncology Group. Phase III trial of ifosfamide with or without paclitaxel in advanced uterine carcinosarcoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Feb 10;25(5):526-31. doi: 10.1200/JCO.2006.06.4907. PMID 17290061
- [Result] Takebayashi Y, Pourquier P, Zimonjic DB, Nakayama K, Emmert S, Ueda T, Urasaki Y, Kanzaki A, Akiyama SI, Popescu N, Kraemer KH, Pommier Y. Antiproliferative activity of ecteinascidin 743 is dependent upon transcription-coupled nucleotide-excision repair. Nat Med. 2001 Aug;7(8):961-6. doi: 10.1038/91008. PMID 11479630
- [Result] Damia G, Silvestri S, Carrassa L, Filiberti L, Faircloth GT, Liberi G, Foiani M, D'Incalci M. Unique pattern of ET-743 activity in different cellular systems with defined deficiencies in DNA-repair pathways. Int J Cancer. 2001 May 15;92(4):583-8. doi: 10.1002/ijc.1221. PMID 11304695
- [Result] Germano G, Frapolli R, Belgiovine C, Anselmo A, Pesce S, Liguori M, Erba E, Uboldi S, Zucchetti M, Pasqualini F, Nebuloni M, van Rooijen N, Mortarini R, Beltrame L, Marchini S, Fuso Nerini I, Sanfilippo R, Casali PG, Pilotti S, Galmarini CM, Anichini A, Mantovani A, D'Incalci M, Allavena P. Role of macrophage targeting in the antitumor activity of trabectedin. Cancer Cell. 2013 Feb 11;23(2):249-62. doi: 10.1016/j.ccr.2013.01.008. PMID 23410977
- [Result] del Campo JM, Sessa C, Krasner CN, Vermorken JB, Colombo N, Kaye S, Gore M, Zintl P, Gomez J, Parekh T, Park YC, McMeekin S. Trabectedin as single agent in relapsed advanced ovarian cancer: results from a retrospective pooled analysis of three phase II trials. Med Oncol. 2013 Mar;30(1):435. doi: 10.1007/s12032-012-0435-1. Epub 2013 Feb 9. PMID 23397080
- [Result] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437